CLINICAL TRIAL: NCT06878963
Title: Comparison of the Effects of Pericapsular Nerve Group Block and Suprainguinal Fascia Iliaca Compartment Block on Neuraxial Anesthesia Positioning and Postoperative Analgesia in Hip Fracture Surgeries
Brief Title: COmparison of PENG Block and SIFICB in Hip Fracture Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Nezir Yılmaz, Associate Professor, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: ADYU-ANS-NY-008
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Hip Fracture; Pericapsular Nerve Group Block (PENG Block); Suprainguinal Fasya Iliaca Block
Keywords: Hip fracture; Pericapsular nerve group block; Suprainguinal fasya iliaca block; Patient positioning
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The researchers performing the nerve block procedures were not involved in the evaluation of the outcomes. Additionally, the researcher responsible for evaluating the outcomes was not involved in the nerve block applications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group P (Experimental): The PENG block will be performed on the patient with the injection of local anesthesia under ultrasound guidance in the femoral region, beneath the biceps tendon.
  Interventions: Procedure: PENG Block
- Group S (Experimental): The SIFIB block will be performed on the patient with the injection of local anesthetic between the iliac fascia and iliac muscle in the femoral region, under ultrasound guidance.
  Interventions: Procedure: SIFICB Block

INTERVENTIONS:
Procedure: PENG Block — The PENG block will be performed on the patient with the injection of local anesthesia under ultrasound guidance in the femoral region, beneath the biceps tendon.
  Arms: Group P
Procedure: SIFICB Block — The SIFIB block will be performed on the patient with the injection of local anesthetic between the iliac fascia and iliac muscle in the femoral region, under ultrasound guidance.
  Arms: Group S

SUMMARY:
The aim of this study is to compare the effectiveness of the PENG block and SIFIB in facilitating the positioning for neuroaxial anesthesia and their impact on the quality of postoperative analgesia.

DETAILED DESCRIPTION:
Hip fractures are a significant health problem that leads to severe morbidity and mortality in elderly individuals. Neuroaxial anesthesia is often preferred in the surgical treatment of these patients due to its ability to maintain hemodynamic stability and manage postoperative analgesia. However, the severe pain accompanying these fractures makes it difficult to achieve an appropriate position for neuroaxial anesthesia, which complicates both patient comfort and the work of the anesthesia provider.

In recent years, peripheral nerve blocks have emerged as an effective method to overcome this challenge. The pericapsular nerve group (PENG) block and supra-inguinal fascia iliaca compartment block (SIFIB) are commonly used techniques for the management of pain related to hip fractures. While studies comparing the analgesic efficacy of these two blocks exist in the literature, data regarding their specific effects on neuroaxial anesthesia positioning are limited.

In this study, patients scheduled for surgery due to hip fractures will receive either a pericapsular nerve group (PENG) block or a supra-inguinal fascia iliaca compartment block (SIFIB). Both block procedures will be performed under ultrasound guidance and sterile conditions, following standard protocols. After the block procedure, the time taken for patients to transition into the neuroaxial anesthesia position (primary outcome) will be measured, and the level of pain experienced during positioning will be assessed using the Visual Analog Scale (VAS).

In the postoperative period, VAS scores and additional analgesic requirements (secondary outcomes) will be recorded for 24 hours. Demographic data (age, gender, body mass index) and comorbidities will also be collected and used for intergroup comparisons. Throughout the study, patient privacy will be respected, and the collected data will be analyzed anonymously.

The study will be conducted in accordance with the Declaration of Helsinki, and informed consent will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Hip fractures
* 40-80 years

Exclusion Criteria:

* Contraindicated to spinal anesthesia
* allergy to local anesthetics
* severe peripheral neuropathy
* mental disorders

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Patient positioning | During neuroaxial block procedure
  In patients with hip fractures, during spinal anesthesia, the angle between the patient's back and the operating table will be recorded while positioning the patient.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) score | During neuroaxial block procedure
  VAS score is a measurement instrument for subjective characteristics of pain. VAS score range from 0 to 10. 0 refers to no pain and 10 refers to the worst pain ever had

IPD SHARING:
Plan to Share IPD: Undecided